CLINICAL TRIAL: NCT04121533
Title: The Influence of Vitamin D Supplementation With and Without Glucosamine Sulfate and Omega-3 Fatty Acids in Patients With Osteoarthritis Symptoms
Brief Title: Vitamin D Supplementation in Knee Osteoarthritis
Acronym: VitD-OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: USANA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1023358
Record Dates: First submitted 2019-10-04; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis, Knee; Vitamin D Supplementation
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Cholecalciferol; Glucosamine; Fatty Acids, Omega-3

STUDY DESIGN:
Intervention Model Description: This study consists of a double-blind, placebo-controlled experimental design. Subjects will be randomly assigned to one of three groups: (#1) vitamin D (cholecalciferol, 4000 IU) with glucosamine sulfate (1000 mg) and omega-3 fatty acids (eicosapentaenoic (EPA, 580 mg) and docosahexaenoic (DHA, 470 mg) acids), (#2) vitamin D (cholecalciferol, 4000 IU) with matching glucosamine sulfate and omega-3 fatty acid placebo supplements, or (#3) matching vitamin D, glucosamine sulfate and omega-3 fatty acid placebo supplements. Supplements will be taken daily for 84 days (12 weeks). Groups will be permuted in random blocks of six.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Matching vitamin D, glucosamine sulfate and omega-3 fatty acid placebo supplements. Supplements taken daily for 84 days (12 weeks).
  Interventions: Dietary Supplement: Placebo
- Vitamin D (Experimental): Vitamin D (cholecalciferol, 4000 IU) with matching glucosamine sulfate and omega-3 fatty acid placebo supplements. Supplements taken daily for 84 days (12 weeks).
  Interventions: Dietary Supplement: Vitamin D (cholecalciferol)
- Vitamin D, glucosamine sulfate, and omega-3 fatty acids (Experimental): Vitamin D (cholecalciferol, 4000 IU) with glucosamine sulfate (1000 mg) and omega-3 fatty acids (eicosapentaenoic (EPA, 580 mg) and docosahexaenoic (DHA, 470 mg) acids). Supplements taken daily for 84 days (12 weeks).
  Interventions: Dietary Supplement: Vitamin D (cholecalciferol); Dietary Supplement: Glucosamine sulfate and omega-3 fatty acids

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo supplement for vitamin D (cholecalciferol), glucosamine sulfate, and omega-3 fatty acids. Supplement was taken orally every day for 84-days.
  Arms: Placebo
Dietary Supplement: Vitamin D (cholecalciferol) — Vitamin D (cholecalciferol). Supplement was taken orally every day for 84-days.
  Arms: Vitamin D; Vitamin D, glucosamine sulfate, and omega-3 fatty acids
Dietary Supplement: Glucosamine sulfate and omega-3 fatty acids — Glucosamine sulfate and omega-3 fatty acids supplement was taken orally every day for 84-days.
  Arms: Vitamin D, glucosamine sulfate, and omega-3 fatty acids

SUMMARY:
Muscular (i.e., quadriceps) weakness is a major risk factor for predisposing the knee to osteoarthritis, impairing physical function, and increasing patient-reported pain. Muscular weakness is a consequence of and could contribute to the development of knee osteoarthritis. Minimizing muscular weakness has been fount to improve activities of daily living in patients with osteoarthritis symptoms. Although vitamin D associates with muscular strength in young and old populations, it is unknown if vitamin D supplementation improves muscular strength in subjects with osteoarthritis or osteoarthritis symptoms. It is also unknown if supplemental vitamin D alters circulating cytokine concentrations in subjects with knee osteoarthritis. Furthermore, it is probable that a more comprehensive supplement is necessary to improve muscular strength. Such as glucosamine sulfate and omega-3 fatty acids (i.e., eicosapentaenoic and docosahexaenoic acids) which could be influential on knee pain and inflammation as well as muscular strength. Therefore, the purpose of this study is to identify the influence of vitamin D supplementation with and without glucosamine sulfate and omega-3 fatty acids on circulating cytokine concentrations and muscular strength in subjects with knee osteoarthritis symptoms. This study is intended to establish preliminary data identifying the influence of vitamin D supplementation on circulating cytokines and muscular strength in subjects with osteoarthritis at no more than minimal risk exposure to subjects.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a degenerative joint condition and a leading contributor to the global burden of disease. Estimates indicate that approximately 14 million people in the United States have symptomatic knee OA, and nearly half of those individuals are between 45 and 65 years of age. Over the years, data have extended our knowledge regarding the early premise of knee OA being the sole consequence of "wear and tear" processes of articular cartilage and it is now recognized that knee OA arises, in part, as a consequence of cytokine-mediated cellular and signaling events.

Cytokines are pleiotropic proteins instrumental to the immune response, host defenses, and intra- and inter-cellular signaling. Tumor necrosis factor (TNF)-α and interleukin (IL)-1β are pro-inflammatory cytokines that promote the catabolic and destructive events of knee OA in animal and human studies. These findings are corroborated by data illustrating chondrocytes as a site for pro-inflammatory cytokine production in knee OA, and that disease severity and progression associate with increasing TNF-α, IL-1β, and other cytokine concentrations in the circulation and transcriptional expression in peripheral blood leukocytes. Fortunately, IL-10 is an anti-inflammatory cytokine expressed in chondrocytes and possesses chondroprotective properties by inhibiting pro-inflammatory cytokine production. While some factors are unavoidable or unpreventable, such as aging, trauma, and genetic predisposition, disrupting the cytokine network could alter OA development and progression.

Low circulating vitamin D concentrations are reported in elderly with and without knee osteoarthritis symptoms. Serum 25(OH)D concentrations associate with muscular strength or performance in elderly. Vitamin D supplementation increases serum 25(OH)D concentrations and improves muscular strength in elderly. Based on these observations, vitamin D is essential for muscle function in elderly, however, it is unknown if supplemental vitamin D influences muscular strength in subjects with knee OA. Furthermore, it is probable that a more comprehensive supplement is necessary to improve muscular strength.

The aim of this study is to identify the influence of supplemental vitamin D on circulating cytokines and muscular strength in subjects with knee OA. This study consists of a double-blind, placebo-controlled experimental design. Subjects will be randomly assigned to one of three groups: (#1) vitamin D (cholecalciferol, 4000 IU) with glucosamine sulfate (1000 mg) and omega-3 fatty acids (eicosapentaenoic (EPA, 580 mg) and docosahexaenoic (DHA, 470 mg) acids), (#2) vitamin D (cholecalciferol, 4000 IU) with matching glucosamine sulfate and omega-3 fatty acid placebo supplements, or (#3) matching vitamin D, glucosamine sulfate and omega-3 fatty acid placebo supplements. Supplements will be taken daily for 84 days (12 weeks). Groups will be permutated in random blocks of six. Serum 25(OH)D, serum cytokines and muscular-based outcomes will be determined prior to, during, and following supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral knee pain, weakness, and impaired physical activity
* Older than 18 years of age but younger than 60 years of age
* Reportedly physically active (minimum of 30 minutes of continuous exercise or physical exertion 3 times per week during the previous year)

Exclusion Criteria:

* Bilateral symptoms of hip, knee or ankle osteoarthritis
* Recent (within 2 years) surgery on the symptomatic or non-symptomatic limb
* History of metabolic bone disease
* History of any skeletal muscle pathologies
* History of cardiac or peripheral cardiovascular system abnormalities
* History of clotting disorders
* History of coronary artery disease, peripheral vascular disease, or stroke
* History of cancer
* Use of warfarin or other anti-coagulants prior to study enrollment
* Use of cholesterol lowering medication
* History of high cholesterol or triglycerides
* History of high blood pressure
* Diagnosed with diabetes mellitus
* Impaired liver function
* Impaired kidney function
* Pregnant
* Daily dietary supplement or vitamin use during the previous year
* Use of corticosteroid medication
* Use of orlistat, phenobarbital, phenytoin, or thiazide
* Morbidly obese (body mass index > 40 kg/m2)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2011-07-28 (Actual); Primary Completion 2013-01-08 (Actual); Study Completion 2013-01-08 (Actual)

PRIMARY OUTCOMES:
Circulating (serum) IL-10 concentration | Day 84
  The influence of supplemental vitamin D on serum IL-10 concentration (pg/mL) in subjects with knee osteoarthritis.
Single-leg peak isokinetic torque | Day 84
  The influence of supplemental vitamin D on single-leg peak isokinetic torque (Nm at 60 degrees per second) in subjects with knee osteoarthritis.

SECONDARY OUTCOMES:
Patient reported pain and physical dysfunction | Day 28 and Day 84
  Patient reported pain and physical dysfunction (using the subsection questions in the WOMAC survey) will be reported by each subject.

OTHER OUTCOMES:
Circulating (serum) cytokines (TNF-alpha, IFN-gamma, IL-2, IL-4, IL-5, IL-6, IL-8, IL-12, IL-13, and IL-1beta) | Day 84
  Supplemental vitamin D influences serum cytokines (pg/mL) in subjects with knee OA
Single leg peak isometric force | Day 84
  Supplemental vitamin D influences single leg peak isometric force (N) in subjects with knee osteoarthritis.
Circulating (serum) soluble cytokine receptors | Day 84
  Supplemental vitamin D influences serum soluble cytokine receptors (sIL-1r, sIL-1r2, sIL-4r, sIL-6r, sTNFr1, and sTNFr2: pg/mL)
Single leg peak power output | Day 84
  Supplemental vitamin D influences single leg peak output (Nm) in subjects with knee osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Barker, PhD, Principal Investigator — Intermountain Health Care, Inc.